CLINICAL TRIAL: NCT03180801
Title: Phase IIb Study of the Efficacy of FLU-v, a Broad Spectrum Influenza Vaccine in an H1N1 Influenza Healthy Human Challenge Model
Brief Title: Efficacy of FLU-v in an H1N1 Influenza Human Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PepTcell Limited (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLU-v-004; 2016-002134-74 (EudraCT Number); 2015-25472 (Other: CRADA between NIAID-NIH and PepTcell)
Record Dates: First submitted 2017-05-31; First posted 2017-06-08 (Actual); Results first posted 2019-05-01 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2019-04

CONDITIONS: Influenza
Keywords: broad; universal; vaccine; influenza; peptide; T cell; H1N1; human challenge
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 adjuvanted placebo (Placebo Comparator): 0.5ml adjuvanted placebo on Day -43 and on Day -22 followed by influenza challenge on day 0
  Interventions: Biological: adjuvanted placebo; Other: Influenza challenge
- Group 2 adjuvanted FLU-v one dose (Experimental): 0.5ml (500mcg) adjuvanted FLU-v vaccine on Day -43 and adjuvanted placebo on Day -22 followed by influenza challenge on day 0
  Interventions: Biological: adjuvanted FLU-v; Biological: adjuvanted placebo; Other: Influenza challenge
- Group 3 adjuvanted FLU-v two doses (Experimental): 0.5ml (500mcg) adjuvanted FLU-v vaccine on Day -43 and on Day -22 followed by influenza challenge on day 0
  Interventions: Biological: adjuvanted FLU-v; Other: Influenza challenge

INTERVENTIONS:
Biological: adjuvanted FLU-v — Subcutaneous injection in the upper arm with 500mcg of FLU-v as 0.5ml emulsion in 0.25ml of WFI and 0.25ml of adjuvant Montanide ISA-51
  Arms: Group 2 adjuvanted FLU-v one dose; Group 3 adjuvanted FLU-v two doses
Biological: adjuvanted placebo — Subcutaneous injection in the upper arm with 0.5ml emulsion made of 0.25ml of WFI and 0.25ml of adjuvant Montanide ISA-51
  Arms: Group 1 adjuvanted placebo; Group 2 adjuvanted FLU-v one dose
Other: Influenza challenge — On day 0, administration with an intranasal sprayer of 1ml of PBS containing 10(7) TCID50 of Influenza A 2009 H1N1 human virus manufactured under GMP in certified Vero cells.

SUMMARY:
FLU-v is a broad spectrum influenza vaccine that targets regions conserved among multiple influenza strains. FLU-v adjuvanted with Montanide ISA-51 was shown to be safe in previous trials. This study aims to assess efficacy of adjuvanted FLU-v vaccine in protecting healthy volunteers against an influenza challenge delivered intranasally under quarantine.

Efficacy of FLU-v will be assessed by measuring the incidence and severity of the disease in the treatment groups compared to the placebo group. In addition, the immune responses of the volunteers to FLU-v will also be explored.

DETAILED DESCRIPTION:
Influenza is a highly variable virus. Most of the variability comes from the proteins on the viral capsid surface; NA and HA. Current vaccines use these highly variable, immunogenic proteins to induce production of neutralising antibodies, however because these proteins are different for each strain, and can also change over time within strains due to antigenic drift, a new vaccine is required each year designed specifically to the strain predicted to circulate that year. In the event of a mismatch between predicted and actual circulating strains, or the emergence of a new strain due to antigenic shift, the effectiveness of the annual vaccine is drastically reduced. These limitations are further compounded by the short manufacturing window between strain prediction and the start of the influenza season, as well as the limited supply of suitable eggs used for vaccine production. As a result of these issues, only a limited supply of annual vaccine is available.

FLU-v, a novel peptide vaccine, aims to provide a broad-spectrum response using peptide antigens matching immunogenic regions of conserved viral proteins found inside the viral capsid. These antigens have been shown to induce cytotoxic T-cell responses and non-neutralising antibodies in both pre-clinical and clinical studies. The FLU-v vaccine administered with and without adjuvant has been demonstrated to be safe in previous trials, and addition of adjuvant Montanide ISA-51 was shown to produce superior immunological responses compared to non-adjuvanted FLU-v. Data from a previous phase IIb study conducted as part of the UNISEC consortium suggest that the cellular and/or humoral responses resulting from vaccination with adjuvanted FLU-v may reduce influenza symptom severity and duration, although the study was not powered to assess these efficacy measures.

Presently, efficacy will be evaluated as a primary endpoint alongside safety as part of a single centre, placebo controlled, phase IIb viral challenge study, using influenza A 2009 H1N1 human virus, in suitable healthy subjects aged 18-60 years. Two dosing regimens will be explored. In addition, immunological endpoints will be addressed as exploratory endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females aged ≥18 and ≤55 years of age at the point of enrolment.
2. Willingness to remain in isolation for the duration of viral shedding and to comply with all study requirements.
3. The following criteria are applicable to subjects in a heterosexual relationship and female subjects in a same sex relationship (i.e., the criteria do not apply to male subjects in a same sex relationship):

   1. True abstinence- when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

      Or
   2. Two forms of effective contraceptive methods among (between) the couple, which are defined as:

      * For males: condom with spermicidal foam/gel/film/cream, sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. This applies only to males participating in the study).
      * For females:

   Women no longer of child bearing potential (post-menopausal females are defined as having a history of amenorrhea for at least 2 years, otherwise they should have documented status as being surgically sterile or post hysterectomy. The latter applies only to females participating in the study). If of childbearing potential, then acceptable forms of contraception include:
   * Established (a minimum of 2 weeks prior to admission) use of oral, injected or implanted hormonal methods of contraception.
   * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
   * Barrier methods of contraception or occlusive cap (diaphragm or cervical/vault caps), both with one of the following - spermicidal foam/gel/film/cream/suppository.

     * The longevity of contraception is as follows:

   Males:
   * Comply with agreed contraception at entry to quarantine, and continuing until 90 days after the date of viral challenge/last dosing with IMP (whichever occurs last).
   * Must not donate sperm following discharge from quarantine until 90 days after the date of viral challenge/last dosing with IMP (whichever occurs last).

   Females:

   If of childbearing potential must have a negative pregnancy test at screening and just prior to the date of Viral Challenge, and must be using contraception consisting of two forms of birth control (one of which must be a barrier method) starting from at least 2 weeks prior to the first vaccination and continuing until 90 days after the date of Viral Challenge/last dosing with IMP (whichever occurs last).
4. Willing to have samples stored for future research.
5. Sero-suitable to the study challenge virus within 90 days of Day 0.
6. Agrees to abstain from alcohol intake 24 hours before admission on Day -2 or Day -1 and all other outpatient visits.
7. Agrees to not use prescription or over-the-counter medications (including aspirin, decongestants, antihistamines, and other NSAIDs), and herbal medication (including, but not limited to, Vitamin C, Vitamin D, immune booster products, herbal tea, St. John's Wort), within 14 days prior to study vaccine administration through the final follow-up visit, unless approved by the investigator and sponsor medical monitor.
8. An informed consent document signed and dated by the subject and the Investigator or delegate.
9. A history of childhood asthma before the age of 12 years is acceptable provided the subject is asymptomatic without treatment. Subjects with a single episode of wheezing (lasting less than 2 weeks) after the age of 12 years can be included at the Investigator's discretion provided the episode was more than 1 year ago and did not require a hospital admission and/or oral/intravenous steroids.
10. In good health with no history of major medical conditions that will interfere with subject safety, as defined by medical history, physical examination, and routine laboratory tests and determined by the Investigator at a screening evaluation.

    * A subject with a history of Herpes type 1 or 2 infection may be included if there are no active lesions present and the subject is not taking active medication.
    * A subject with or without any evidence of atopy including any history of allergic rhinitis, dermatitis, and conjunctivitis will be included as long as they do not conflict with exclusion criteria. Mild to moderate arthritis of non-inflammatory origin may be allowed if the subject is not at risk from relative immobility in the Quarantine Unit and does not require regular medication.
11. A documented medical history for a minimum of the last 2 years prior to inoculation.

Exclusion Criteria:

1. Any subjects who have smoked 10 pack years at any time. Of those subjects that have smoked less than 10 pack years at any time, a subject will be excluded: If regular smokers (e.g., smoking every day) at the time of enrolment. If current casual smoker or use of smoking / nicotine-related products, they must agree to refrain from smoking during the in-patient stay
2. Presence of self-reported or medically documented significant medical condition including but not limited to:

   * Chronic pulmonary disease (e.g., asthma (except what is stated in inclusion criteria 9), COPD)
   * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
   * Chronic medical conditions requiring close medical follow-up or hospitalisation during the past 5 years (e.g., insulin dependent diabetes mellitus, renal dysfunction, haemoglobinopathies).
   * Immunosuppression, or immunodeficiency or ongoing malignancy.
   * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
   * Post infectious or post vaccine neurological sequelae.
   * Hyperlipidemia requiring medical therapy per current American College of Cardiology (ACC) and American Heart Association (AHA) guidelines published in 2013.
3. Individual with body mass index (BMI) <18 and >35.
4. Acute illness within 7 days of first vaccine administration day
5. Clinically significant abnormal electrocardiogram (ECG) and/or parameters, as determined by the Investigator
6. Subjects with clinically significant abnormal systolic and diastolic blood pressure or clinically significant abnormal pulse rate.
7. Subject has abnormal pulmonary function as measured by spirometry defined as a forced vital capacity or forced expiratory volume in 1 second (FEV1) < 80% of predicted or peripheral arterial oxygen saturation (SpO2) < 92% on room air.
8. Known allergy to treatments for influenza (including but not limited to oseltamivir, nonsteroidals).
9. Known allergy to 2 or more classes of antibiotics (e.g. penicillins, cephalosporins, fluoroquinolones, or glycopeptides). Known allergy to excipients in the challenge virus inoculum
10. Daily or household contact with vulnerable populations.
11. Receipt of any investigational drug:

    * within 3 months prior to the planned date of Viral Challenge/first dosing with IMP (whichever occurs first).
    * Receipt of three or more investigational drugs within the previous 12 months prior to the planned date of Viral Challenge/first dosing with IMP (whichever occurs first).
    * Prior inoculation with a virus from the same virus-family as the Challenge Virus.
    * Prior participation in another Human Viral Challenge study with a respiratory virus in the preceding 12 months taken from the date of Viral Challenge/first dosing with IMP (whichever occurs first) in the previous study to the date of expected Viral Challenge in this study.
12. Receipt of any vaccine within 6 months of enrolment.
13. Self-reported or known history of alcoholism or drug abuse (including marijuana) within 6 months prior to enrolment, or positive urine/serum test for drugs of abuse during the study
14. Self-reported or known history of psychiatric or psychological issues that require treatment and are deemed by the PI to be a contraindication to protocol participation.
15. History of a previous severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis.
16. History or evidence of autoimmune disease or known immunodeficiency of any cause - with the exception of atopic dermatitis/eczema and atopic rhinitis.
17. Subjects with any history of physician diagnosed and/or objective test confirmed asthma (except as per inclusion criteria 9), reactive airway disease, COPD, pulmonary hypertension, or chronic lung condition of any aetiology.
18. Positive human immunodeficiency virus (HIV) within 60 days of first vaccination visit, active hepatitis A (HAV), B (HBV), or C (HCV) test.
19. Any significant abnormality altering the anatomy of the nose or nasopharynx (including significant nasal polyps).
20. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
21. Any nasal or sinus surgery within 6 months of Viral Challenge.
22. Recurrent history of fainting.
23. Those employed or immediate relatives of those employed at hVIVO or the Sponsor.
24. Any clinically significant history of epistaxis (nosebleeds) within the last 12 months and/or history of being hospitalized due to epistaxis on any previous occasion.
25. Females who:

    * Are breastfeeding,
    * or have been pregnant within 6 months prior to the study,
    * or have a positive pregnancy test at any point during screening or prior to first dosing with IMP.
26. Presence of fever, defined as subject presenting with a temperature reading of > 38.0°C on Day -43
27. Receipt of blood or blood products, or loss (including blood donations) of 470 mL or more of blood during the 3 months prior to the planned date of first dosing with IMP or planned during the 3 months after the final visit.
28. Receipt of systemic (intravenous and/or oral) glucocorticoids or systemic antiviral drugs within 6 months prior to the planned date of first dosing with IMP.
29. Any other finding that, in the opinion of the Investigator, deems the subject unsuitable for the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Dennison, Dr, Principal Investigator — Hammersmith Medicines Research; Balpreet Matharu, Dr, Principal Investigator — hVIVO Services Limited; Matthew J Memoli, M.D, Study Director — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- hVIVO Services Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoloff GA, Caparros-Wanderley W. Synthetic multi-epitope peptides identified in silico induce protective immunity against multiple influenza serotypes. Eur J Immunol. 2007 Sep;37(9):2441-9. doi: 10.1002/eji.200737254. PMID 17668898
- [Background] Pleguezuelos O, Robinson S, Stoloff GA, Caparros-Wanderley W. Synthetic Influenza vaccine (FLU-v) stimulates cell mediated immunity in a double-blind, randomised, placebo-controlled Phase I trial. Vaccine. 2012 Jun 29;30(31):4655-60. doi: 10.1016/j.vaccine.2012.04.089. Epub 2012 May 8. PMID 22575166
- [Background] Pleguezuelos O, Robinson S, Fernandez A, Stoloff GA, Mann A, Gilbert A, Balaratnam G, Wilkinson T, Lambkin-Williams R, Oxford J, Caparros-Wanderley W. A Synthetic Influenza Virus Vaccine Induces a Cellular Immune Response That Correlates with Reduction in Symptomatology and Virus Shedding in a Randomized Phase Ib Live-Virus Challenge in Humans. Clin Vaccine Immunol. 2015 Jul;22(7):828-35. doi: 10.1128/CVI.00098-15. Epub 2015 May 20. PMID 25994549
- [Background] Pleguezuelos O, Robinson S, Fernandez A, Stoloff GA, Caparros-Wanderley W. Meta-Analysis and Potential Role of Preexisting Heterosubtypic Cellular Immunity Based on Variations in Disease Severity Outcomes for Influenza Live Viral Challenges in Humans. Clin Vaccine Immunol. 2015 Aug;22(8):949-56. doi: 10.1128/CVI.00101-15. Epub 2015 Jun 17. PMID 26084515
- [Background] van Doorn E, Pleguezuelos O, Liu H, Fernandez A, Bannister R, Stoloff G, Oftung F, Norley S, Huckriede A, Frijlink HW, Hak E. Evaluation of the immunogenicity and safety of different doses and formulations of a broad spectrum influenza vaccine (FLU-v) developed by SEEK: study protocol for a single-center, randomized, double-blind and placebo-controlled clinical phase IIb trial. BMC Infect Dis. 2017 Apr 4;17(1):241. doi: 10.1186/s12879-017-2341-9. PMID 28376743
- [Background] Memoli MJ, Czajkowski L, Reed S, Athota R, Bristol T, Proudfoot K, Fargis S, Stein M, Dunfee RL, Shaw PA, Davey RT, Taubenberger JK. Validation of the wild-type influenza A human challenge model H1N1pdMIST: an A(H1N1)pdm09 dose-finding investigational new drug study. Clin Infect Dis. 2015 Mar 1;60(5):693-702. doi: 10.1093/cid/ciu924. Epub 2014 Nov 20. PMID 25416753
- [Derived] Ponne S, Kumar R, Vanmathi SM, Brilhante RSN, Kumar CR. Reverse engineering protection: A comprehensive survey of reverse vaccinology-based vaccines targeting viral pathogens. Vaccine. 2024 Apr 11;42(10):2503-2518. doi: 10.1016/j.vaccine.2024.02.087. Epub 2024 Mar 23. PMID 38523003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An excess number of subjects were vaccinated to ensure 123 subjects were able to complete the quarantine period . Any subject that dropped out after vaccination but before inoculation with the challenge virus was replaced with another vaccinated subject.
Groups:
- Group 1 Adjuvanted Placebo: 0.5ml adjuvanted placebo (Montanide ISA-51: WFI) on Day -43 and on Day -22 as subcutaneous injection followed by H1N1 influenza challenge on day 0.
- Group 2 Adjuvanted FLU-v One Dose: 0.5ml (500mcg) adjuvanted FLU-v vaccine on Day -43 and adjuvanted placebo on Day -22 as subcutaneous injection followed by H1N1 influenza challenge on day 0.
- Group 3 Adjuvanted FLU-v Two Doses: 0.5ml (500mcg) adjuvanted FLU-v vaccine on Day -43 and on Day -22 as subcutaneous injection followed by H1N1 influenza challenge on day 0.
Period: Overall Study
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Started | 50 | 52 | 51
Safety Population (The safety population included all vaccinated subjects) | 50 | 52 | 51
Intention to Treat (ITT included all vaccinated and inoculated subjects) | 42 | 40 | 41
Completed | 42 | 40 | 41
Not Completed | 8 | 12 | 10
Not completed — Physician Decision | 3 | 3 | 1
Not completed — Non-compliance | 1 | 4 | 0
Not completed — Inoculation Target Reached | 1 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: The Intention to treat (ITT) group was used for all analysis. ITT includes those participants who received both vaccination and challenge with an influenza virus.
Groups:
- Group 1 Adjuvanted Placebo: adjuvanted placebo on Day -43 and on Day -22 followed
- Group 2 Adjuvanted FLU-v One Dose: 500mcg adjuvanted FLU-v vaccine on Day -43 and adjuvanted placebo on Day -22
- Group 3 Adjuvanted FLU-v Two Doses: 500mcg adjuvanted FLU-v vaccine on Day -43 and on Day -22
- Total: Total of all reporting groups
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses | Total
Number analyzed (Participants) | 42 | 40 | 41 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (7.5) | 29.9 (8.9) | 27.4 (9.2) | 28.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 11 | 36
  Male | 29 | 28 | 30 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 33 | 37 | 34 | 104
  Ethnicity: Asian/Asian British | 1 | 0 | 1 | 2
  Ethnicity: Black/Black British | 3 | 0 | 2 | 5
  Ethnicity: Chinese | 0 | 1 | 0 | 1
  Ethnicity: Hispanic | 0 | 1 | 0 | 1
  Ethnicity: Japanese | 1 | 0 | 0 | 1
  Ethnicity: Mixed | 4 | 0 | 3 | 7
  Ethnicity: Other | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 42 | 40 | 41 | 123
Number of subjects with challenge strain HAI titers > or = 40 at screening [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mild to Moderate Influenza Disease (MMID)
Description: To determine the effect of FLU-v on reducing the incidence of Mild to Moderate Influenza Disease (MMID) defined as detectable viral shedding by Luminex Respiratory Pathogen Panel Test (RPP) in the presence of at least one influenza symptom.
Time Frame: From 24h post-viral inoculation (Day 1) until the end of the quarantine phase on Day 7
Population: ITT includes those participants who received both vaccination and were challenged with the H1N1 influenza virus
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 Adjuvanted Placebo: 0.5ml adjuvanted placebo on Day -43 and on Day -22
- Group 2 Adjuvanted FLU-v One Dose: 0.5ml (500mcg) adjuvanted FLU-v vaccine on Day -43 and adjuvanted placebo on Day -22
- Group 3 Adjuvanted FLU-v Two Doses: 0.5ml (500mcg) adjuvanted FLU-v vaccine on Day -43 and on Day -22
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 42 | 40 | 41
Participants
  positive MMID | 23 | 13 | 15
  Negative MMID | 19 | 27 | 26
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Fisher exact test is used to test if vaccine group has lower MMID rate than placebo; Test type: Other; p = 0.03, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Fisher exact test is used to test if vaccine group has lower MMID rate than placebo; Test type: Other; p = 0.07, Fisher Exact

2. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) Per Subject.
Description: To determine the number of TEAEs that were reported after the first administration of the vaccine until the end of the study (overall) and then separated into pre-inoculation (events reported from the time of first vaccination up to Day 0 prior to time of inoculation) and post-inoculation (Day 0 inoculation time through study completion).
Time Frame: From the first vaccination on day -43 to the last follow up visit on day 63.
Population: Safety population
Measure: Mean (Standard Error); unit: Number of TEAEs per subject
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 50 | 52 | 51
Number of TEAEs per subject
  Overall | 1.86 (0.26) | 1.38 (0.24) | 2.35 (0.27)
  Pre-inoculation | 1.00 (0.21) | 0.81 (0.13) | 1.51 (0.19)
  Post-Inoculation | 0.86 (0.16) | 0.58 (0.15) | 0.84 (0.16)
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One sided Fisher's exact test is used to test if the TEAE rates pre-inoculation recorded for the treatment group are higher than for placebo; Test type: Other — One sided Fisher's exact test is used to test if TEAE rates of vaccine group is higher than the placebo group; p = 0.647, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Fisher's exact test is used to test if TEAE rate of vaccine group recorded pre-inoculation is higher than placebo; Test type: Other; p = 1.00, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One sided Fisher's exact test is used to test if TEAE rate of vaccine group post-inoculation is higher than the placebo group; Test type: Other; p = 0.0240, Fisher Exact
Statistical Analysis 4: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.186, Fisher Exact

3. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Event Classified by Relatedness and Severity.
Description: Number of subjects with one or more AE are reported by severity (mild, moderate and severe) and relatedness to vaccine or challenge virus inoculation (definitely, probably, possibly, unlikely, not related).
Time Frame: From the day of the first vaccination up to the end of the study on day +63.
Population: Safety population
Measure: Number; unit: Number of participants
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 50 | 52 | 51
Number of participants
  Subjects with TEAEs definately related to vaccine | 7 | 24 | 29
  Subjects withTEAEs probably related to vaccine | 1 | 0 | 6
  Subjects with TEAEs possibly related to vaccine | 3 | 2 | 3
  Subjects with TEAEs unlikely related to vaccine | 11 | 4 | 9
  Subjects with TEAEs not related to vaccine | 37 | 21 | 34
  Subjects with TEAEs definately related to virus | 1 | 0 | 0
  Subjects with TEAEs probably related to virus | 3 | 1 | 1
  Subjects with TEAEs possibly related to virus | 4 | 3 | 6
  Subjects with TEAEs unlikely related to virus | 7 | 0 | 6
  Subjects with TEAEs not related to virus | 37 | 32 | 44
  Subjects with mild TEAEs | 37 | 33 | 42
  Subjects with moderate TEAEs | 13 | 4 | 11
  Subjects with Severe TEAEs | 0 | 1 | 3
  Subjects with Serious Adverse Events (SAEs) | 0 | 0 | 0

4. Secondary Outcome: Number of Subjects With Detectable Viral Shedding and Number of Subjects With Recorded Influenza Symptoms During the Quarantine Period.
Description: Number of subjects experiencing at least one influenza symptom and at least two influenza symptoms.
  Number of subjects with detectable shedding by RPP (Luminex) test from nasal swabs.
  Number asymptomatic subjects with detectable virus by RPP (Luminex) test from nasal swabs.
Time Frame: Quarantine period from day 1 to day 7 post-inoculation.
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 42 | 40 | 41
Participants
  Subjects with at least one symptom | 37 | 34 | 30
  Subjects with at least two symptoms | 27 | 16 | 23
  Subjects with detectable shedding | 23 | 15 | 18
  Asymptomatic subjects with detectable shedding | 0 | 2 | 3
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Fisher exact test is used to test if vaccine group has lower rate of subjects experiencing at least one symptom; Test type: Other; p = 0.465, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.074, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Fisher exact test is used to test if vaccine group has lower rate of subjects experiencing at least two symptoms; Test type: Other; p = 0.024, Fisher Exact
Statistical Analysis 4: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; [analysis description as in outcome 4, analysis 3]; Test type: Other; p = 0.230, Fisher Exact
Statistical Analysis 5: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Fisher exact test is used to test if vaccine group has lower rate of subjects with detectable virus shedding; Test type: Other; p = 0.09, Fisher Exact
Statistical Analysis 6: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Fisher exact test is used to test if vaccine group has lower rate of subjects with detectable virus shedding; Test type: Other; p = 0.22, Fisher Exact
Statistical Analysis 7: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Fisher exact test is used to test if vaccine group has lower rate of subjects asymptomatic with detectable virus shedding; Test type: Other; p = 0.23, Fisher Exact
Statistical Analysis 8: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; [analysis description as in outcome 4, analysis 7]; Test type: Other; p = 0.12, Fisher Exact

5. Secondary Outcome: Viral Shedding Duration
Description: Number of days with detectable viral shedding measured using the Luminex Respiratory Pathogen Panel test.
Time Frame: starting from evening of Day 1 post-inoculation up to Day 7.
Population: ITT
Measure: Mean (Standard Error); unit: days
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 42 | 40 | 41
days | 1.95 (0.36) | 1.20 (0.31) | 1.90 (0.39)
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Wilcoxon test is used to test if vaccine group has shorter shedding duration than placebo; Test type: Other; p = 0.0501, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Wilcoxon test is used to test if vaccine group has shorter shedding duration than placebo; Test type: Other; p = 0.3139, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Total Viral Shedding (Area Under the Curve)
Description: Shedding is quantified by RT-PCR from nasal swabs taken twice daily (am/pm) during the quarantine period. Plotting the log copy number/ml for each time point against time is done to calculate the area under the curve (AUC) using the trapezoidal rule.
Time Frame: from the evening of Day 1 post-inoculation to the morning of Day 7 (last timepoint before expected quarantine discharge)
Population: ITT
Measure: Mean (Standard Error); unit: hours*log10copy number/ml
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 42 | 40 | 41
hours*log10copy number/ml | 153.67 (33.39) | 98.47 (27.39) | 138.79 (31.73)
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Wilcoxon test is used to test if vaccine group has smaller shedding AUC than placebo; Test type: Other; p = 0.102, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Wilcoxon test is used to test if vaccine group has a smaller shedding AUC than placebo; Test type: Other; p = 0.481, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Peak Viral Load
Description: Shedding is quantified by RT-PCR from nasal swabs taken twice daily (am/pm) during the quarantine period. Peak viral load is the highest recorded log10copy number/ml.
Time Frame: as for outcome 6
Population: ITT
Measure: Mean (Standard Error); unit: log10copy number/ml
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 42 | 40 | 41
log10copy number/ml | 2.24 (0.40) | 1.54 (0.39) | 2.28 (0.42)
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Wilcoxon test is used to test if vaccine group has lower peak viral shedding than placebo; Test type: Other; p = 0.128, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Wilcoxon test is used to test if vaccine group has lower peak viral shedding than placebo; Test type: Other; p = 0.601, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Duration of Influenza Symptoms
Description: Subjects were assessed by the physician whilst under quarantine post-inoculation. The number of days subjects experienced influenza symptoms was recorded.
Time Frame: as for outcome 6
Population: ITT
Measure: Mean (Standard Error); unit: days
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 42 | 40 | 41
days | 3.26 (0.37) | 2.67 (0.35) | 2.76 (0.37)
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Wilcoxon test is used to test if vaccine group has shorter duration of symptoms than placebo; Test type: Other; p = 0.142, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Wilcoxon test is used to test if vaccine group has shorter duration of symptoms than placebo; Test type: Other; p = 0.147, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Number of Symptoms Experienced Per Subject Per Day.
Description: Mean of total number of symptoms (upper and lower respiratory and systemic symptoms) experienced calculated as the total sum of symptoms experienced divided by the number of days in which symptoms were collected.
Time Frame: from the evening of Day 1 post-inoculation to the morning until the day of last symptom noted during the expected quarantine period (up tp Day 7)
Population: ITT
Measure: Mean (Standard Error); unit: number of symptoms per day
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 42 | 40 | 41
number of symptoms per day | 2.57 (0.33) | 2.08 (0.32) | 2.51 (0.41)
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Wilcoxon test is used to test if vaccine group has fewer average number of symptoms than placebo; Test type: Other; p = 0.080, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Wilcoxon test is used to test if vaccine group has fewer average number of symptoms than placebo; Test type: Other; p = 0.271, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Peak Number of Symptoms Experienced Per Subject in a Single Day.
Description: The highest level of the total sum of all upper and lower respiratory tract and systemic symptoms recorded on any day starting from the evening of Day 1 post-inoculation until the day of last symptom noted during the expected quarantine period (up to Day 7).
Time Frame: from the evening of Day 1 post-inoculation until the day of last symptom noted during the expected quarantine period (up to Day 7).
Population: ITT
Measure: Mean (Standard Error); unit: number of symptoms
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 42 | 40 | 41
number of symptoms | 2.12 (0.26) | 1.68 (0.22) | 1.88 (0.28)
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Wilcoxon test is used to test if vaccine group has fewer peak symptoms than placebo; Test type: Other; p = 0.099, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Wilcoxon test is used to test if vaccine group has fewer peak symptoms than placebo; Test type: Other; p = 0.178, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Assessment of Self-reported Influenza Symptoms by FLU-PRO Questionnaire.
Description: FLU-PRO assesses 32 influenza symptoms. Subjects rate each symptom on a 5-point ordinal scale, with higher scores indicating a more frequent sign or symptom. For 27 of the items, the scale is as follows: 0 ("Not at all"), 1 ("A little bit"), 2 ("Somewhat"), 3 ("Quite a bit"), and 4 ("Very much"). For 5 items, severity is assessed in terms of numerical frequency, i.e., vomiting or diarrhea (0 times, 1 time, 2 times, 3 times, or 4 or more times); with frequency of sneezing, coughing, and coughed up mucus or phlegm evaluated on a scale from 0 ("Never") to 4 ("Always").The FLU-PRO total score is computed as a mean score across all 32 items comprising the instrument. Total scores can range from 0 (symptom free) to 4 (very severe symptoms).
Time Frame: from Day 1 post-inoculation until the day 7.
Population: ITT
Measure: Mean (Standard Error); unit: FLU-PRO total score
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 42 | 40 | 41
FLU-PRO total score | 0.05 (0.01) | 0.03 (0.01) | 0.04 (0.01)
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; One-sided Wilcoxon test is used to test if vaccine group has lower FLU-PRO scores than placebo; Test type: Other; p = 0.064, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; One-sided Wilcoxon test is used to test if vaccine group has lower FLU-PRO scores than placebo; Test type: Other; p = 0.201, Wilcoxon (Mann-Whitney)

12. Other Pre Specified Outcome: Immunogenicity of FLU-v
Description: To determine the antibody responses specific to FLU-v.
Time Frame: At pre-inoculation post-vaccination (Day -2), and post-influenza challenge (Day 35/Day 63)
Population: Subjects that received vaccination, underwent influenza challenge and provided serum samples.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
Number analyzed (Participants) | 41 | 40 | 40
ng/ml
  Day -2 | 5.94 (0.99) | 72.17 (6.28) | 75.74 (5.50)
  Day 35 | 6.09 (0.93) | 66.86 (6.07) | 73.55 (5.69)
  Day 63 | 6.26 (1.06) | 60.33 (5.81) | 67.90 (5.35)
Statistical Analysis 1: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; comparison on day -2; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; Comparion on day -2; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; Comparison on day 35; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; Comparison on day 35; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 5: Comparison: Group 1 Adjuvanted Placebo vs Group 2 Adjuvanted FLU-v One Dose; Comparison on day 63; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 6: Comparison: Group 1 Adjuvanted Placebo vs Group 3 Adjuvanted FLU-v Two Doses; Comparison on day 63; Test type: Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the date of first administration of vaccine to the date of inoculation with the challenge virus (TEAEs).
Description: Treatment Emergent AEs are all AEs that occur in the period between the first administration of the vaccine and the end of the study independently of their intensity and if they are related or not to the vaccine.
Arm/Group | Group 1 Adjuvanted Placebo | Group 2 Adjuvanted FLU-v One Dose | Group 3 Adjuvanted FLU-v Two Doses
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 27/50 | 33/52 | 45/51
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Adjuvanted Placebo (N=50) | Group 2 Adjuvanted FLU-v One Dose (N=52) | Group 3 Adjuvanted FLU-v Two Doses (N=51)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Injection site induration (General disorders) | 9 (9) | 24 (24) | 31 (31)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (6) | 0 (0) | 3 (3)
Oral Herpes (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 9 (9) | 8 (8)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 11 (11) | 5 (5) | 13 (13)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI requires the Sponsor's consent to publish any material that contains Sponsor Property; including Study Data.

DOCUMENTS (3):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT03180801/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03180801/SAP_001.pdf
  • Informed Consent Form (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT03180801/ICF_002.pdf